CLINICAL TRIAL: NCT03823313
Title: Feasibility, Acceptability and Preliminary Effects of the Spiritual Care Assessment and Intervention (SCAI) Framework for Adults With Advanced Cancer and Their Caregivers (FCGs): A Clinical Pilot Trial
Brief Title: Feasibility, Acceptability and Preliminary Effects of the Spiritual Care Assessment and Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Indiana University Health (Other)
Responsible Party: Principal Investigator, Alexia M. Torke, Associate Professor of Medicine and Associate Division Chief of General Internal Medicine and Geriatrics, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IUSCC-0665
Record Dates: First submitted 2019-01-29; First posted 2019-01-30 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Advanced Cancer; Metastatic Cancer
Keywords: Spiritual Care; Religion; Spirituality; Caregiver
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spiritual Care Assessment and Intervention (Experimental)
  Interventions: Behavioral: SCAI (Spiritual Care Assessment and Intervention)

INTERVENTIONS:
Behavioral: SCAI (Spiritual Care Assessment and Intervention) — 4 sessions completed with an IU Health chaplain using a framework of questions called the Spiritual Care Assessment And Intervention tool. The weekly sessions will focus on one of the 4 areas of spiritual experience (meaning and purpose, relationships, transcendence and peace, self-worth and identity)

SUMMARY:
The purpose of this study is to test a spiritual care intervention for adults with advanced cancer and their caregivers. This intervention will assess 4 areas of spiritual experience: meaning and purpose, relationships, transcendence and peace, self-worth and identity. Participants will be asked to complete questionnaires and participate in 4 sessions with research chaplains.

DETAILED DESCRIPTION:
Several studies have shown that cancer affects multiple dimensions of a patient's life as well as the lives of caregivers and others close to the patient who, when faced with life crises, may use religion and spirituality (R/S) to cope. This study is the first of its kind to incorporate a semi-structured spiritual care and intervention (SCAI) framework into the spiritual care of advanced cancer patients while maintaining proper controls in order to investigate its feasibility, acceptability and potential effects on the emotional and spiritual outcomes of advanced cancer patients and their caregivers. This framework will assess 4 areas of spiritual experience: meaning and purpose, relationships, transcendence and peace, self-worth and identity. Additionally, not only will this study assess acceptability and feasibility of the intervention, it will also track and document coping, satisfaction, anxiety, depression, quality of life outcomes and follow-up with both patient and caregivers following Spiritual Care Assessment and Intervention (SCAI).

Specific Aim 1: To evaluate the feasibility and acceptability of the SCAI intervention for adults with advanced cancer and their caregivers.

Specific Aim 2: To establish our ability to collect outcome data to support a future efficacy trial for patients and their caregivers in the outpatient clinic and home setting.

Specific Aim 3: To test the preliminary impact of the SCAI intervention on patient and caregiver spiritual wellbeing (primary outcome) and quality of life, religious coping, depression, and anxiety (secondary outcomes)

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age.
* Patient is at least 2 weeks post-diagnosis of an incurable and advanced stage (IV) lung, colorectal, GI neuroendocrine and Hepatobiliary, testicular and esophageal solid malignancy and receiving cancer care at IU Simon Cancer Center.
* Patient is willing and able to consent, has a reliable phone and willing to participate in 4 sessions of 30 (+/- 5) minutes per session.
* Patient has a family member or eligible friend considered to be a caregiver and interested in participating in the study.
* Patient has adequate English fluency for completion of data collection.
* Family Caregiver (FCG) is at least 18 years of age.
* Family Caregiver (FCG) has been invited to participate in the trial with a patient who meets eligibility criteria above.
* Family Caregiver (FCG) is willing and able to consent and to participate in 4 sessions of 30 (+/- 5) minutes per session
* Family Caregiver (FCG) has adequate English fluency for completion of data collection.

Exclusion Criteria:

* Patient makes 3 or more errors on a validated 6-item cognitive screener (Appendix A) or exhibits significant psychiatric or cognitive impairment (e.g., dementia/delirium, retardation, active psychosis) that in the judgment of the investigators would preclude providing informed consent and study participation.
* Currently receiving hospice care (patients who enroll in hospice during the trial will have the option of continuing trial participation).
* Family Caregiver (FCG) exhibits significant psychiatric or cognitive impairment (e.g., dementia/delirium, retardation, active psychosis) that in the judgment of the investigators would preclude providing informed consent and study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Rate of enrollment | from recruitment to enrollment (i.e. up to 30 days)
  number of eligible patients that are consented and enrolled in the trial
Attendance Rate | 4 weeks
  proportion of participants who attend all four intervention sessions
Mean Satisfaction Score | 4 weeks
  satisfaction score among participants on the satisfaction survey
Functional assessment of chronic illness therapy-Spiritual Well-being Scale Scores | baseline, 1-2 weeks after session 4, 6 weeks, 3 months
  Total score at baseline will be compared to score at to the score at 1 week, 6 weeks, and 3 months

SECONDARY OUTCOMES:
Percentage of completed baseline surveys | baseline
  percentage of completed baseline surveys in enrolled patients
Percentage of completed follow up surveys | baseline, 1-2 weeks after session 4, 6 weeks, 3 months
McGrill Quality of Life Questionnaire score | baseline, 1-2 weeks after session 4, 6 weeks, 3 months
  Measure of patient quality of life through total score at baseline compared to score at 1 week, 6 weeks, and 3 months
Caregiver Quality of Life Index-Cancer Questionnaire score | baseline, 1 week, 6 weeks, 3 months
  Measure of caregiver quality of life through total score at baseline compared to score at 1 week, 6 weeks, and 3 months
Caregiver Quality of Life Index-Cancer Questionnaire score | baseline, 1-2 weeks after session 4, 6 weeks, 3 months
  Measure of caregiver quality of life through total score at baseline compared to score at 1 week, 6 weeks, and 3 months
Generalized Anxiety Disorder Scale Scores | baseline, 1-2 weeks after session 4, 6 weeks, 3 months
  Measure of Anxiety through total score at baseline compared to score at 1 week, 6 weeks, and 3 months
Patient Health Questionnaire Depression Scale (PHQ-8) | baseline, 1 week, 6 weeks, 3 months
  Measure of depression through total score at baseline compared to score at 1 week, 6 weeks, and 3 months
Brief RCOPE score | baseline, 1-2 weeks after session 4, 6 weeks, 3 months
  Measure of coping through total score at baseline compared to score at 1 week, 6 weeks, and 3 months
Intervention Satisfaction Questionnaire score | baseline, 1-2 weeks after session 4, 6 weeks, 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexia Torke, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Melvin & Bren Simon Cancer Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No